CLINICAL TRIAL: NCT06741384
Title: Effect of Breathing Exercises on Depression and Sexual Function in Postmenopausal Women
Brief Title: Breathing Exercises on Depression in Postmenopausal Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Middle East University (Other)
Responsible Party: Principal Investigator, Saher Lotfy El Gayar, Assistant Professor of Physical Therapy, Middle East University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Breathing Exercises
Record Dates: First submitted 2024-12-17; First posted 2024-12-19 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Postmenopausal; Depressive Symptom; Breathing Exercises
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diaphragmatic breathing exercises group (Active Comparator): 30 women participating in diaphragmatic breathing plus aerobic training.
  Interventions: Other: Diaphragmatic breathing exercises; Other: Aerobic training
- Control group (Active Comparator): 30 women participating in aerobic training only.
  Interventions: Other: Aerobic training

INTERVENTIONS:
Other: Diaphragmatic breathing exercises — Participants will be directed to position their hands on the rectus abdominis muscle located under the anterior chest wall while resting in a hook position. They will be instructed to inhale slowly and deeply via the nostrils, expanding their abdomen without raising their upper chest, and resting their shoulders. Following the cessation of respiration, the woman will slowly exhale by pursing her lips. A respiratory cycle will consist of a three-second inhalation, a three-second pause, and a six-second exhalation. The diaphragmatic training regimen will consist of doing 3-5 sets of 5-10 deep breaths, with 2-minute intervals of rest in between sets.
  Arms: Diaphragmatic breathing exercises group
Other: Aerobic training — The women will participate in aerobic training on cycle ergometer. Each session will consist of 30-45 minutes of cycling at a moderate intensity, accompanied by a workout heart rate ranging from 65% to 75% of the maximal heart rate and ranging between 12 and 14 on the Borg rating of perceived exertion 20-point scale. After ten minutes of warm-up, every session will end with a brief 3-minute period of cool-down.

SUMMARY:
Evaluate the effect of breathing exercises on depression and sexual function in postmenopausal women

DETAILED DESCRIPTION:
Sixty postmenopausal women will be sourced from the Obstetrics & Gynecology outpatient clinic at El Mahalla El Kobra general hospital in Egypt, with referrals from gynecologists. Patients will be randomly assigned into two groups.

Study group: It will include 30 women participating in diaphragmatic breathing plus aerobic training.

Control group: It will include 30 women participating in aerobic training.

At baseline and poststudy, the following outcomes will be assessed:

1. Depression (Beck Depression Inventory II scale).
2. Sexual function (female sexual function index questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* Minimum of 3 years after menopause.
* Mild to moderate depression.
* Mild to moderate sexual dysfunction.
* Their ages will be ranged from 45 to 60 years old.
* Their BMI will be less than 30 kg/m2.

Exclusion Criteria:

* Prolapse of the pelvic organs.
* Pelvic tumors.
* Vaginal infections.
* Musculoskeletal/ neurological limitations to exercise.
* Psychiatric disorders.
* Unstable cardiovascular conditions.
* Diabetes.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females
Enrollment: 60 (Estimated)
Dates: Start 2024-12-26 (Estimated); Primary Completion 2025-03-20 (Estimated); Study Completion 2025-03-25 (Estimated)

PRIMARY OUTCOMES:
Depression | At baseline and after 8 weeks
  The second edition of Beck depression inventory scale will be scored. The second edition of Beck depression inventory scale consists of 21- items. Item scores ranging from 0 to 3 are combined to produce a total score that ranges from 0 to 63 using the cumulative scoring technique. Elevated scores suggest a more severe level of depression.

SECONDARY OUTCOMES:
Sexual function | At baseline and after 8 weeks
  Female sexual function index questionnaire will be scored. The female sexual function index questionnaire is a 19-item, self-report measure of female sexual function that provides scores on overall levels of sexual function. The 19 items of the female sexual function index questionnaire use a 5-point scale ranging from 1 to 5 with higher scores indicating greater levels of sexual functioning on the respective item. Total scores of 26.5 or lower characterize sexual dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Sayed Saif, Ph.D, Study Director — National institute for Gerontology

IPD SHARING:
Plan to Share IPD: No